CLINICAL TRIAL: NCT06017934
Title: PIVOT Trial: Promoting Increased Physical Activity in Hospitalised Older Adults With Trained Volunteers: An Implementation Feasibility Study
Brief Title: Promoting Increased Physical Activity in Hospitalised Older Adults
Acronym: PIVOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Leeds (Other); Portsmouth Hospitals NHS Trust (Other Government); Salisbury NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Frimley Park Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ERGO 84163
Record Dates: First submitted 2023-07-18; First posted 2023-08-30 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hospital-associated Deconditioning
Keywords: Physical activity; Hospital-associated deconditioning; Sedentary behaviour; Physical inactivity; Volunteer-led; Feasibility; Implementation
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care
- Volunteer-led physical activity (Experimental): Trained volunteers will deliver walking, or bedside exercises with hospitalised older adults twice per day.
  Interventions: Behavioral: Volunteer-led physical activity

INTERVENTIONS:
Behavioral: Volunteer-led physical activity — Participants will be assessed by the therapy team who will prescribe tailored activity and then liaise with the mobility volunteers, who will deliver the intervention. Participants who can mobilise independently will be encouraged to perform walking exercises, progressing their walking distance over set markers in the hospital (e.g., to the end of the bed and back; to the doorway and back; to the toilet and back). Participants who require assistance in mobility will perform bed (e.g., hip abduction, static quads), or chair exercises (e.g., ankle pumps, knee extension, arm raise), and will be progressed to performing walking exercises when their physical function improves. Volunteers will check with nursing staff that participants are safe to exercise before each activity session. Participants will receive the mobility sessions twice daily, starting upon recruitment and continuing until the day of discharge from hospital.
  Arms: Volunteer-led physical activity

SUMMARY:
The PIVOT study will explore the feasibility of training volunteers to deliver exercise to hospitalised older adults to improve the health of older people and prevent deconditioning while in hospital. Loss of strength and mobility (i.e., deconditioning) is common in hospitalised older people and is associated with a decline in physical function, poorer quality of life and increased health and care costs. Physical inactivity is an important and modifiable risk factor. A previous study showed it is feasible to train volunteers to engage with older people in hospital and facilitate walking and bedside exercises. The intervention was well-received by older adults, staff members and volunteers. The aim of this study is to determine the feasibility of implementing volunteer-led physical activity in three hospitals of varying sizes in different regions.

Older adults aged 65 years and above admitted to an acute hospital will be invited to participate in the study. The study aims to recruit 180 participants; 90 from three intervention sites and 90 from a control site. Participants at the intervention sites will receive a twice daily volunteer-led physical activity intervention, and participants at the control site will receive usual care.

Participants who are able to mobilise independently will perform walking exercises and individuals with mobility impairments will perform bedside exercises. The volunteers will be trained and monitored by hospital therapists. The acceptability of the intervention will be explored through interviews with patients, volunteers, and staff. Intervention feasibility will also be examined through measuring retention of trainers, volunteers, and patients on the intervention, and adherence to the exercise.

Study findings will help to determine the feasibility of the volunteer-led physical activity intervention across different sized hospitals, voluntary service teams, and therapy services to explore the implementation and roll out of the intervention across NHS sites and the development of a toolkit to support knowledge transfer.

DETAILED DESCRIPTION:
Aim The aim of the current research is to explore whether volunteers can be trained to deliver exercise support to older adults across three different sized hospitals in different locations. Researchers will also explore if the intervention is accepted by patients, volunteers and staff and if it has any benefits on patients' health and functional outcomes (e.g., quality of life and muscle strength).

Study Design This is a multicentre feasibility study using mixed methods (i.e., quantitative and qualitative measures) to explore the implementation of a volunteer-led physical activity intervention to older adults in hospital. The study will include three intervention sites and one control site. Feasibility studies are used to determine whether an intervention is appropriate for further evaluation, to determine sample sizes for controlled trials and to assess whether the ideas and findings can be shaped to be relevant and sustainable.

Sample Size A sample size of 180 patients, 90 intervention (30 from each intervention site) and 90 from the control site, was chosen in line with previous sample size recommendations for feasibility studies of 24-50 participants. This sample size was considered an appropriate number that is pragmatic and achievable within the study timescale and resources available at each site.

This research aims to recruit 15 volunteers at each site to provide sufficient cover to deliver the intervention. In a previous study (SoMoVe trial) 17 volunteers were recruited, 16 completed training and 12 were retained.

Recruitment and Consent Older adults with an acute medical admission to four hospitals will be screened for eligibility by research nurses. Eligible patients will be introduced to the study by ward staff. Those who are interested in the study will be approached by the research team for further information and information sheets will be provided. Written informed consent will be obtained from all patients who agree to participate in the study.

Volunteers will be invited by hospital voluntary services within each hospital site. The voluntary services team will send the interested volunteers details to the research team, who will then get in contact to complete informed consent.

Inclusion and Exclusion Criteria Patients: The inclusion criteria are adults aged 65 years and above who are able to provide informed consent. Exclusion criteria are anyone with a severe cognitive impairment (MoCA less than 10), patients isolated for infection control reasons, and patients receiving end of life care.

Volunteers: The inclusion criteria for volunteers are age 18 years and above, who have completed the generic clearance and training with the hospital voluntary services, who can provide written informed consent, and are able to communicate fluently enough in English. Fluent English is required to ensure the intervention content can be delivered clearly and thus safely to participants. Volunteers that are unable to safely complete the exercises included in the intervention will be excluded from the study.

Intervention The exercises were developed based on clinical expertise from therapists and from our previous research of volunteer-led mobility interventions in hospital (SoMoVe study). Participants will be assessed by the therapy team who will prescribe tailored activity and then liaise with the mobility volunteers, who will deliver the intervention. Participants who can mobilise independently will be encouraged to perform walking exercises, progressing their walking distance over set markers in the hospital (e.g., to the end of the bed and back; to the doorway and back; to the toilet and back). Participants who require assistance in mobility will perform bed (e.g., hip abduction, static quads), or chair exercises (e.g., ankle pumps, knee extension, arm raise), and will be progressed to performing walking exercises when their physical function improves. Volunteers will check with nursing staff that participants are safe to exercise before each activity session. Participants will receive the mobility sessions twice daily, starting upon recruitment and continuing until the day of discharge from hospital.

Training The volunteer training package was developed by a clinician and therapist and will cover topics including patient and personal safety, mobility and exercise training, and response to adverse evets, such as falls. Volunteers will participate in practical sessions to practice the exercises with peers. When ready, volunteers will work with patients, initially under close supervision and when deemed competent by the trainer, they will be encouraged to support mobility sessions independently. A volunteer competency checklist will be completed and signed off by the trainer before volunteers work independently. The training will be delivered by a physiotherapist in each intervention site.

Fidelity Checks Throughout the study period, fidelity checks will be conducted by the trainers once every 2 weeks to ensure that the volunteers are delivering high quality and safe exercise. The volunteers will be observed and assessed against a competency and implementation checklist, including personal safety, basic patient safety, pre-intervention tasks (e.g., safe set up of exercise space), and exercise delivery (e.g., showing safe and effective exercise technique). Volunteers will be asked to keep an attendance record during the intervention using session completion logs. Regular monthly volunteer meetings will be scheduled online to discuss experiences and gain feedback from peers and trainers. Based upon fidelity checks and volunteer feedback, extra one-to-one training sessions will be available if necessary. The principle investigator will also visit intervention sites to observe and liaise with volunteers and trainers.

Data Collection Data including age, sex, co-morbidities, medications, functional status, and cognition will provide participants' baseline characteristics in both intervention and control sites.

Volunteer data including age, occupation, qualifications, volunteering experience, any physiotherapy, sport or therapeutic experience, and employment status will be collected. Data on the study sites including hospital size, size of voluntary service team, the number of hospital volunteers, and information on the therapy services and what usual care looks like will be collected to provide contextual information.

The primary outcome measures are feasibility (can it be done?) and acceptability (will volunteers, staff, and patients accept and embrace the programme?) of the intervention.

Feasibility will be assessed by:

1. Number of trainers trained and retained in each hospital site (total number and %)
2. Number of volunteers recruited, trained, and retained (total number and %)
3. Recruitment rate (%) of participants in each site
4. Adherence to the intervention (total number and %)

Acceptability will be assessed through process evaluation involving:

1. Observation and monitoring of volunteer training
2. Interviews with therapy managers to establish usual care in each site
3. Observation of the interaction between volunteers, patients, and healthcare professionals on the wards, including contextual factors that may potentially influence the delivery and receipt of the intervention.

Qualitative interviews will be conducted with service managers, therapy managers, patients, nurses, ward therapists, and volunteers from all study sites, to determine the acceptability of the intervention. Purposive sampling will be conducted to capture a range of experiences and opinions from patients of varying age and mobility levels, staff with varying seniority and gender mix, and volunteers with a range of volunteering experience, age groups, and gender mix. The interviews will explore barriers and facilitators to the implementation of the intervention into routine clinical practice.

Fidelity Assessment Fidelity assessment will be conducted across all study sites to ensure that the exercises and prescribed dose are delivered by the volunteers as prescribed. Volunteers will be trained to document each physical activity session in participant exercise diaries, detailing whether all the exercises were carried out as prescribed, or whether some exercises were excluded, and reasons for exclusions. The exercise diaries will be affixed to participants' activity prescription sheet. Further assessments of fidelity of volunteer training and the intervention will be conducted through site visits by the research fellow once every 2 months and to address any issues that arise.

Secondary Outcome Measures The secondary outcome measures will include assessment of physical activity levels (StepWatch Activity Monitor; SAM; Modus health, Washington, USA), physical function (Short Physical Performance Battery and grip strength), and quality of life (EuroQol; EQ-5D-5L). Moreover, data on length of hospital stay and hospital readmission will be accessed through electronic patient records. Data collection will be conducted by research nurses, supported by the local principal investigators.

Data Analysis Primary Outcome Analyses Participants' baseline characteristics will be described using summary statistics, including mean (standard deviations), medians (interquartile ranges), counts and proportions, as appropriate. Statistical analysis will be conducted using the statistical software SPSS. Summary statistics will be used to describe the feasibility of recruiting, training, and retaining the trainers, the volunteers and study participants. Participants' exercise diaries will be analysed to determine how many physical activity sessions were offered and the number and percentage of completed sessions.

Data collected from the interviews will be transcribed verbatim and analysed using thematic analysis (TA). The audio- recordings will be transcribed by an administrative colleague within the research department who is experienced in transcribing qualitative data. TA is a method for identifying, analysing and reporting patterns or themes within data and is widely used in qualitative research. Transcribed text will be read and coded separately and then together by two researchers. The codes will be analysed to generate concepts and ideas to determine the acceptability of the intervention, and to identify facilitators and barriers to the implementation process. The codes act as tags or labels to help catalogue key concepts embedded within the raw data. From the codes, themes will be developed to reflect the views and experiences of the older adults and volunteers regarding the volunteer-led physical activity intervention.

Secondary Outcome Analyses Daily step count, Short Physical Performance Battery, grip strength, and quality of life measured on recruitment and discharge, and length of hospital stay will be analysed as continuous variables. The completion rate of each data item will be measured. The distribution of each outcome measure will be assessed for normality and described using parametric or non-parametric statistics accordingly. Hospital readmission in 3 and 6 months will be analysed as a categorical variable. Where there is missing data, the main analyses will be based on available data.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Adults aged 65 years and above
* Able to provide written informed consent

Volunteers

* Adults aged 18 years and above
* Completed the generic clearance and training with the hospital voluntary services
* Able to provide written informed consent
* Able to communicate fluently enough in English. Fluent English is required to ensure the intervention content can be delivered clearly and thus safely to participants.

Exclusion Criteria:

Patients

* Anyone with a severe cognitive impairment (MoCA less than 10)
* Patients isolated for infection control reasons
* Patients receiving end of life care

Volunteers

* Volunteers that are unable to safely complete the exercises included in the intervention will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview data exploring the acceptability of the intervention, including barriers and enablers to the implementation of the intervention. | through intervention completion, an average of 2 months
  Qualitative interviews will be conducted with service managers, therapy managers, patients, nurses, ward therapists, and volunteers from all study sites, to determine the acceptability of the intervention.
The number of volunteers recruited to the study (%). | through study completion, an average of 3 years
  Feasibility of recruiting volunteers to deliver the physical activity intervention at each hospital site
Number of trainers trained in each hospital site (%) | through study completion, an average of 3 years
  Feasibility of recruiting therapists to deliver the intervention at each hospital site.
Adherence to the intervention (%) | through study completion, an average of 3 years
  The number of participants retained in the intervention at each hospital site.
Recruitment rate (%) of participants in each site | through study completion, an average of 3 years
  Feasibility of recruiting older adults onto the volunteer-led physical activity intervention at each hospital site.
The number of volunteers trained at the end of the study period (%) | through study completion, an average of 3 years
  Feasibility of training volunteers to deliver the physical activity intervention at each hospital site
The number of volunteers retained at the end of the study period (%) | through study completion, an average of 3 years
  Feasibility of retaining volunteers to deliver the physical activity intervention at each hospital site
Number of trainers retained in each hospital site (%) | through study completion, an average of 3 years
  Feasibility of retaining therapists to deliver the intervention at each hospital site.

SECONDARY OUTCOMES:
Patient's subjective assessment of quality of life - visual analogue scale (VAS) | Baseline and post intervention, an average of 2 months
  Quality of life will be measured using the EuroQol (EQ-5D-5L) VAS. The VAS subjectively rates health from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Grip strength | Baseline and post intervention, an average of 2 months
  Grip strength is a simple and accurate measure of muscle function in clinical practice. Grip strength will be measured using the Jamar hand dynamometer, the most widely used instrument in clinical practice with established test-retest, inter-rater and intra-rater reliability.
Short Physical Performance Battery (SPPB) | Baseline and post intervention, an average of 2 months
  The SPPB is a reliable and valid measure of physical function in older people ≥ 60 years and includes exploration of three domains, including walking speed, chair stands, and three progressive balance tasks.
Physical activity | 7 days upon recruitment
  Physical activity will be measured using the StepWatch Activity Monitor (SAM; Modus health, Washington, USA), recording daily step count. The SAM is worn on the ankle and is considered an accurate measure of physical activity in older hospitalised patients that engage in low-intensity physical activity and have lower walking speeds.
Patient's subjective assessment of quality of life - EuroQol (EQ-5D-5L) | Baseline and post intervention, an average of 2 months
  Quality of life will be measured using the EuroQol (EQ-5D-5L) assessment comprising a short descriptive questionnaire. The questionnaire includes 5 domains (e.g., mobility; self-care; usual activities; pain/discomfort; and anxiety/depression) measured with 5 response levels from 'no problems' to 'extreme problems/unable'.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Frimley Park Hospital, Frimley, Surrey
  - Salisbury District Hospital, Salisbury, Wiltshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim S, Ibrahim K, Dodds R, Purkis A, Baxter M, Rogers A, Sayer AA, Roberts HC. Physical activity in hospitalised older people: the feasibility and acceptability of a volunteer-led mobility intervention in the SoMoVe study. Age Ageing. 2020 Feb 27;49(2):283-291. doi: 10.1093/ageing/afz114. PMID 31566671
- [Background] Meredith SJ, Roberts H, Grocott MPW, Jack S, Murphy J, Varkonyi-Sepp J, Bates A, Lim SER. Frail2Fit study protocol: a feasibility and acceptability study of a virtual multimodal intervention delivered by volunteers to improve functional outcomes in older adults with frailty after discharge from hospital. BMJ Open. 2023 Mar 16;13(3):e069533. doi: 10.1136/bmjopen-2022-069533. PMID 36927597
- [Background] Lim SER, Meredith S, Agnew S, Clift E, Ibrahim K, Roberts H. Evaluating the feasibility and acceptability of virtual group exercise for older adults delivered by trained volunteers: the ImPACt study protocol. BMJ Open. 2022 Feb 1;12(2):e052631. doi: 10.1136/bmjopen-2021-052631. PMID 35105576